CLINICAL TRIAL: NCT05568875
Title: Happy Hands - an E-self-management Intervention for People With Hand Osteoarthritis
Acronym: HappyHands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Dam Foundation (Other)
Responsible Party: Principal Investigator, Anne Therese Tveter, Professor, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 477746
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-04

CONDITIONS: Hand Osteoarthritis
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial with a qualitative study nested within the trial
Who Masked: Investigator
Masking Description: Only investigator conduction the analyses will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-self-management intervention (Experimental): 12-week e-self-management intervention consisting of exercise videos and videos with information about recommended treatment
  Interventions: Other: e-self-management intervention (Happy Hands app); Other: Treatment as usual
- Treatment as usual (Active Comparator): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: e-self-management intervention (Happy Hands app) — The 12-week intervention consists of 30 short informational videos addressing the themes prioritized by the patient research partners. These themes are further operationalized into the following categories: "Information on hand OA", "Hand exercises", "Use of assistive devices and orthoses", "Medication and surgical alternatives", and "Self-management of the disease". Additionally, the intervention includes a hand exercise program consisting of 8 videos providing instructions on warm up, exercises to improve mobility, strength and coordination, and a stretching exercise. The intervention group will additionally receive treatment as usual.
  Arms: e-self-management intervention
Other: Treatment as usual — Treatment as usual may vary from no treatment at all to referral to a patient education group program, or occupational therapy.

SUMMARY:
The main aim of this project is to assess the effect, cost-effectiveness and user experiences with using an e-self-management intervention in addition to treatment as usual compared to treatment as usual alone in patients with hand osteoarthritis. The study is an RCT comprising approx 400 participants with hand osteoarthritis recruited from primary and secondary healthcare in all four health regions in Norway.

DETAILED DESCRIPTION:
Hand osteoarthritis (OA) is a highly prevalent rheumatic joint disease, and the number of people living with debilitating hand OA will continue to rise in the coming decades due to increased life expectancy. Research shows that patients with hand OA have poor access to recommended treatment, and in Norway, they are increasingly referred to surgical consultation before having received recommended first-line treatment. Thus, there is a need to develop easily viable models of care for patients with hand OA that make recommended treatment available across different healthcare levels.

Our hypotheses are that an e-self-management intervention for people with hand OA will improve pain and function and be more cost-effective compared to treatment as usual, and that this app can easily be implemented in both specialist and primary healthcare. The hypotheses will be tested and explored in a randomized controlled trial, with a qualitative study nested within this trial.

The main research questions are:

1. To evaluate whether a 12-week e-self-management intervention is more effective in improving pain and function (according to the OMERACT-OARSI responder criteria26) compared to usual care in patients with hand OA (randomized controlled trial).
2. To determine the cost-effectiveness of the e-self-management intervention compared to usual care after 6 months (randomized controlled trial).
3. To explore patients' experience of barriers and facilitators for adopted and continued use of a e-self-management intervention for treatment of hand OA (qualitative interviews).

Secondary research questions will also be assessed.

Approx 400 patients will be recruited in this multicenter randomized controlled trial where patients with hand OA are allocated to either usual care or a 12-week e-self-management intervention delivered through a smartphone app (the HAPPY Hands app). Outcome measures are collected at baseline, 3 months (=end of intervention) and 6 months

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with hand osteoarthritis
* Possessing a smartphone

Exclusion Criteria:

* cognitive deficits
* are scheduled for hand surgery within the next 3 months
* do not talk or understand Norwegian,
* have uncontrolled serious comorbidities

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Most women
Enrollment: 386 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
OMERACT/OARSI responder criteria | Baseline and 3 months follow-up
  Combined score of change in pain, function and disease activity. Patients are categorized into responders or non-responders according to the following:
  High improvement on pain or function:
  1. ≥50% improvement + absolute change of ≥2 in pain (numeric rating scale, NRS 0-10), OR
  2. ≥50% improvement + absolute change of ≥0.6 in function (Measure of Activity Performance of the Hand, MAP-Hand)
  Improvement in at least two of the three following:
  1. ≥20% improvement + absolute change of ≥1 in pain (NRS)
  2. ≥20% improvement + absolute change of ≥0.3 in function (MAP-Hand)
  3. ≥20% improvement + absolute change of ≥1 in global assessment of disease activity (NRS)

SECONDARY OUTCOMES:
OMERACT/OARSI responder criteria long-term | 3 and 6 months follow-up
  Combined score of change in pain, function and disease activity. Patients are categorized into responders or non-responders according to the following:
  High improvement on pain or function:
  1. ≥50% improvement + absolute change of ≥2 in pain (numeric rating scale, NRS 0-10), OR
  2. ≥50% improvement + absolute change of ≥0.6 in function (Measure of Activity Performance of the Hand, MAP-Hand)
  Improvement in at least two of the three following:
  1. ≥20% improvement + absolute change of ≥1 in pain (NRS)
  2. ≥20% improvement + absolute change of ≥0.3 in function (MAP-Hand)
  3. ≥20% improvement + absolute change of ≥1 in global assessment of disease activity (NRS)
Pain intensity | Baseline, 3 and 6 months follow-up
  Numeric rating scale (0-10), 0=no pain, 10= worst possible pain
Pain intensity (intervention group) | 3 times weekly in the intervention period (12 weeks)
  Numeric rating scale (0-10), 0=no pain, 10= worst possible pain, measured after each exercise session
Stiffness | Baseline, 3 and 6 months follow-up
  Numeric rating scale (0-10),0=no stiffness, 10= worst possible stiffness
Stiffness (intervention group) | 3 times weekly in the intervention period (12 weeks)
  Numeric rating scale (0-10),0=no stiffness, 10= worst possible stiffness, measured after each exercise session
Disease activity | Baseline, 3 and 6 months follow-up
  Numeric rating scale (0-10), 0=no disease activity; 10=high disease activity
Disease activity (intervention group) | Monthly in the intervention period (12 weeks)
  Numeric rating scale (0-10), 0=no disease activity; 10=high disease activity, measured each month in the intervention period
Measure of Activity performance (MAP-Hand) | Baseline, 3 and 6 months follow-up
  18 questions conserning activity performance of the hand (1=no problem, 4=cannot do the activity), mean score from 1-4.
Measure of Activity performance (MAP-Hand) (intervention group) | Monthly in the intervention period (12 weeks)
  18 questions conserning activity performance of the hand (1=no problem, 4=cannot do the activity), mean score from 1-4.
Grip strength | Baseline and 3 months follow-up
  Measured with Jamar dynamometer (kg), mean of two measures for each hand
Quality indicators for hand osteoarthritis treatment | Baseline, 3 and 6 months follow-up
  Quality indicators based on the OA-QI questionnaire, adopted to fit the treatment recommendations of hand osteoarthritis. 16 questions answered with yes, no or not appriopriate/do not know. Measured as pass rate.
eHealth literacy | Baseline
  Measured with the eHEALS questionnaire, Norwegian version. 8 questions conserning eHealth literacy (strongly disagree - strongly agree)
Number of painful joints | Baseline
  Number of painful joints on left and right hand
Change in condition | Baseline, 3 and 6 months follow-up
  Global rating of change scale, likert scale with 7 answer options from much better to much worse
Change in condition (intervention group) | Monthly in the intervention group (3 months)
  Global rating of change scale, likert scale with 7 answer options from much better to much worse
Motivation for hand exercises | Baseline and 3 monhts follow-up
  Numeric rating scale (0-10), 0=no motivation, 10=best motivation
Health-related quality of life | Baseline, 3 and 6 months follow-up
  Measured with EQ5D-5L, 5 questions used to calculate an utility score (0-1, 1= best health), assessed as a total score across all timepoints
Health care utilization | Baseline, 3 and 6 months follow-up
  Costs related to self-reported healthcare use in primary and secondary health care. Patients will be asked if they have been seeking healthcare (yes/no), if yes, they will be asked to specify type of healthcare use and time used.
Medication use | Baseline, 3 and 6 months follow-up
  Medication use will be self-reported by the patient
Adverse events | 3 and 6 months follow-up
  Number of adverse events, serious adverse events, and withdrawals because of adverse events. Will be self-reported
Sickleave | Baseline, 3 and 6 months follow-up
  Sickleave due to hand osteoarthritis will be self-reported
Fatigue | Baseline, 3 and 6 months follow-up
  Fatigue last week measured on an 11-point NRS (0=no fatigue, 10=worst possible fatigue)
Patient satisfaction with care | Baseline, 3 and 6 months follow-up
  1 item with five point response options ranging from "Very satisfied" to "Very dissatisfied", higher value indicate better outcome
System Usability Scale (SUS) | 3 month follow-up
  Questionnaire assessing the usability of the Happy Hands app, 10 questions (strongly agree - strongly disagree), index from 0-100 where 100 is best score
Adherence to exercise | 3 times weekly during the intervention period (3 months)
  Number of exercises performed (0-36 exercise sessions), collected from the app
Adherence to exercise long-term | 3 and 6 months follow-up
  Number of exercises performed after completion of intervention, collected from the app
Adherence to informational videos | During the intervention period (3 months)
  Number of informational videos watched, collected from the app
Adherence to informational videos long-term | 3 and 6 months follow-up
  Number of informational videos watched, collected from the app
Arthritis self-efficacy scale | Baseline
  Measured by Arthritis Self-Efficacy Scale (ASES): comprises 11 items addressing pain and symptoms (scored on a 5-point scale ranging from not confident at all to very confident). The scores are summed up to a 0-100 score where higher score indicate better self-efficacy.
Demographic variable | Baseline
  Age, gender, other painful joints, sivil status, education, previous hand surgery, previous treatment, comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Anne Therese Tveter, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (19):
- Norway (19):
  - Arendal sykehus, Arendal
  - Ålesund sjukehus, Ålesund
  - Haukeland Universitetssykehus, Bergen
  - Aurskog Fysikalske Institutt, Bjørkelangen
  - Nordlandssykehuset, Bodø
  - Lærdal Sjukehus, Førde
  - Finnmarkssykehuset, Kirkenes Sykehus, Kirkenes
  - Kongsvinger sykehus, Kongsvinger
  - Kristiansand sykehus, Kristiansand
  - Levanger sykehus, Levanger
  - Revmatismesykehuset Lillehammer, Lillehammer
  - Meråker kurbad, Meråker
  - Nøtterøy Fysioterapi, Nøtterøy
  - Diakonhjemmet Hospital, Oslo
  - Humana Helse, Sandvika
  - Universitetssykehuset Nord-Norge, Tromsø
  - St.Olavs Hospital, Trondheim
  - Helsehuset Stokke, Tønsberg
  - Vikersund bad, Vikersund

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data be made available when upon reasonable request to the principal investigator. The data are not available before they can be anonymoused.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol will be available from 1.11.22. SAP will be available before initation of analyses.
Access Criteria: E-mail the principal investigator for access to supporting information.

REFERENCES:
- [Derived] Fjeldstad KA, Tveter AT, Rasmussen E, Olden L, Nyheim S, Blanck T, Killingmo RM, Kjeken I. Changing Habits With the Happy Hands App: Qualitative Focus Group Study of a Hand Osteoarthritis Self-Management Intervention. J Med Internet Res. 2026 Feb 2;28:e82773. doi: 10.2196/82773. PMID 41628446
- [Derived] Tveter AT, Fjeldstad KA, Varsi C, Maarnes MK, Pedersen SJ, Christensen BS, Blanck T, Nyheim SB, Prior Y, Bjork M, Pelle T, Kjeken I. Evaluation of an e-self-management intervention (Happy Hands app) for hand osteoarthritis: Study protocol for a multicentre randomised controlled trial. Rheumatol Int. 2025 Jan 16;45(1):30. doi: 10.1007/s00296-025-05787-6. PMID 39820549

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT05568875/SAP_000.pdf